CLINICAL TRIAL: NCT06819488
Title: A Clinical Study of Mass Balance of [14C]HRS-7535 in Healthy Adult Chinese Subjects
Brief Title: A Clinical Study of Mass Balance of [14C]HRS-7535
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7535-106
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]HRS-7535 (Experimental)
  Interventions: Drug: [14C]HRS-7535

INTERVENTIONS:
Drug: [14C]HRS-7535 — [14C]HRS-7535.

SUMMARY:
The objective is to evaluate the mass balance of [14C]HRS-7535 in healthy adult Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily sign the informed consent form (ICF) prior to any activities related to the study, demonstrate understanding of the study procedures and methods, and commit to strictly adhering to the clinical trial protocol to complete the study.
2. Healthy male subjects aged between 18 and 45 years (inclusive), determined at the time of signing the informed consent.
3. Male subjects must weigh ≥ 50 kg and have a body mass index (BMI) between 19 and 26 kg/m² (inclusive).
4. Male subjects with female partners of childbearing potential must have no plans for procreation or sperm donation from the time of signing the informed consent until one year after the last dose of the study drug. They must also agree to use highly effective contraception methods (including their partners) during this period.

Exclusion Criteria:

1. Subjects with abnormalities identified through a comprehensive physical examination, vital signs assessment, laboratory tests, chest X-ray, 12-lead ECG, or abdominal ultrasound that are deemed clinically significant by the investigator.
2. Subjects with QTcF ≥ 450 msec at screening or baseline, or any other abnormalities considered clinically significant by the investigator.
3. Subjects who test positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antigen/antibody combination, or syphilis-specific antibodies.
4. Subjects with a history of drug abuse, drug dependence (based on medical history), or those who test positive for drug abuse during urine screening prior to dosing.
5. Subjects who have used any prescription drugs, over-the-counter medications, herbal medicines, or dietary supplements within 2 weeks prior to screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
The time of maximum observed concentration (Tmax) | 0-120 hours.
The maximum observed concentration (Cmax) | 0-120 hours.
The terminal half-life (t1/2) | 0-120 hours.
The total body clearance for extravascular administration (CL/F) | 0-120 hours.
The total radioactivity ratio for blood | 0-96 hours.
The total radioactivity ratio for plasma | 0-96 hours.

SECONDARY OUTCOMES:
Adverse events (AEs) | 0-11 days.
Serious adverse events (AEs) | 0-11 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided